CLINICAL TRIAL: NCT05429073
Title: A Phase 1, Double-Blind, Placebo-Controlled, Single Ascending Dose Study in Healthy Volunteers to Evaluate the Safety, Tolerability, and Pharmacokinetics of RGLS8429
Brief Title: A Study of RGLS8429 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regulus Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: RGLS8429-01
Record Dates: First submitted 2022-05-26; First posted 2022-06-23 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
Keywords: RGLS8429; Autosomal Dominant Polycystic Kidney Disease; ADPKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This will be a double-blinded, randomized, placebo-controlled study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- RGLS8429, first dose level (Experimental): Eligible participants will receive subcutaneous injection of the first dose level RGLS8429 or placebo
  Interventions: Drug: RGLS8429; Drug: Placebo volume-matching RGLS8429 dose
- RGLS8429, second dose level (Experimental): Eligible participants will receive subcutaneous injection of the second dose level RGLS8429 or placebo
  Interventions: Drug: RGLS8429; Drug: Placebo volume-matching RGLS8429 dose
- RGLS8429, third dose level (Experimental): Eligible participants will receive subcutaneous injection of the third dose level RGLS8429 or placebo
  Interventions: Drug: RGLS8429; Drug: Placebo volume-matching RGLS8429 dose
- RGLS8429, fourth dose level (Experimental): Eligible participants will receive subcutaneous injection of the fourth dose level RGLS8429 or placebo
  Interventions: Drug: RGLS8429; Drug: Placebo volume-matching RGLS8429 dose

INTERVENTIONS:
Drug: RGLS8429 — solution for subcutaneous injection
Drug: Placebo volume-matching RGLS8429 dose — solution for subcutaneous injection

SUMMARY:
Primary Objective

• To assess the safety and tolerability of single ascending doses of RGLS8429

Secondary Objectives

* To identify dose-limiting toxicity (DLT) and to determine the maximum tolerated dose (MTD) of a single SC dose of RGLS8429
* To characterize the pharmacokinetic (PK) properties of RGLS8429

DETAILED DESCRIPTION:
In this randomized, double-blind, placebo-controlled Phase 1 study, a single ascending dose of RGLS8429 or placebo will be administered via subcutaneous (SC) injection to healthy volunteers to evaluate the safety, tolerability, and PK of RGLS8429.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 55 years of age
2. Body mass index (BMI) 18 to 35 kg/m2
3. Medically healthy, with no clinically significant medical history in the opinion of the Investigator
4. Estimated glomerular filtration rate (eGFR) ≥ 90 mL/min/1.73 m2
5. Must understand and consent to the study procedures explained in the informed consent form (ICF) and be willing and able to comply with the protocol

Exclusion Criteria:

1. Subject is mentally incapacitated or has significant emotional problems
2. Any medical condition or social circumstance that, in the opinion of the Investigator, may make the subject unlikely to complete the study or comply with study procedures and requirements, or may pose a risk to the subject's safety
3. History or presence of alcoholism or drug abuse within the past 2 years prior to Screening
4. Participation in another clinical trial and/or exposure to any investigational drug or approved therapy for investigational use within 28 days or 5 half-lives of the investigational drug's dosing, whichever is longer, prior to dosing. The 28-day and 5-half-life windows will be calculated from the date of the last dosing in the previous study to Day 1 of the current study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rekha Garg, MD, Study Director — Regulus Therapeutics
Locations (1):
- ICON Early Phase Services, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- RGLS8429, First Dose Level: Eligible participants will receive subcutaneous injection of the first dose level RGLS8429.
  RGLS8429: solution for subcutaneous injection
- RGLS8429, Second Dose Level: Eligible participants will receive subcutaneous injection of the second dose level RGLS8429.
  RGLS8429: solution for subcutaneous injection
- RGLS8429, Third Dose Level: Eligible participants will receive subcutaneous injection of the third dose level RGLS8429.
  RGLS8429: solution for subcutaneous injection
- RGLS8429, Fourth Dose Level: Eligible participants will receive subcutaneous injection of the fourth dose level RGLS8429.
  RGLS8429: solution for subcutaneous injection
- Matching Placebo: Eligible participants will receive subcutaneous injection of the placebo volume-matching RGLS8429 dose.
  Placebo volume-matching RGLS8429 dose: solution for subcutaneous injection
Period: Overall Study
Arm/Group | RGLS8429, First Dose Level | RGLS8429, Second Dose Level | RGLS8429, Third Dose Level | RGLS8429, Fourth Dose Level | Matching Placebo
Started | 6 | 6 | 6 | 6 | 8
Completed | 6 | 6 | 6 | 6 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RGLS8429, First Dose Level | RGLS8429, Second Dose Level | RGLS8429, Third Dose Level | RGLS8429, Fourth Dose Level | Matching Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 8 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.3 (9.48) | 33.8 (6.68) | 34.2 (6.18) | 38.2 (9.28) | 43.9 (6.58) | 37.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5 | 2 | 8 | 20
  Male | 3 | 4 | 1 | 4 | 0 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 5 | 2 | 7 | 24
  Not Hispanic or Latino | 0 | 2 | 1 | 4 | 1 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 2 | 0 | 1 | 5
  White | 6 | 4 | 4 | 5 | 7 | 26
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events (AEs)
Description: Incidence and severity of adverse events after administration of RGLS8429
Time Frame: Baseline to Day 29
Population: Safety Population: all subjects who received a dose of study drug; subjects were analyzed based on treatment received
Measure: Number; unit: participants
Arm/Group | RGLS8429, First Dose Level | RGLS8429, Second Dose Level | RGLS8429, Third Dose Level | RGLS8429, Fourth Dose Level | Matching Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
participants
  Number of subjects with Grade 3, 4 or 5 treatment-emergent adverse events | 0 | 0 | 0 | 0 | 0
  Number of subjects with Treatment-emergent adverse events leading to discontinuation | 0 | 0 | 0 | 0 | 0
  Number of Subjects with Serious Adverse Events or deaths | 0 | 0 | 0 | 0 | 0
  Number of subjects with at least one treatment-emergent adverse event | 1 | 1 | 3 | 1 | 3

2. Secondary Outcome: Incidence of DLT and Determination of MTD
Description: Identify dose limiting toxicity and the maximum tolerated dose after RGLS8429 administration
Time Frame: Baseline to Day 29
Reporting Status: Not Posted

3. Secondary Outcome: Plasma Half-life (T1/2) of RGLS8429
Description: Measure plasma elimination half-life after RGLS8429 administration
Time Frame: Baseline to Day 15
Reporting Status: Not Posted

4. Secondary Outcome: Plasma Clearance of RGLS8429
Description: Measure plasma clearance after RGLS8429 administration
Time Frame: Baseline to Day 15
Reporting Status: Not Posted

5. Secondary Outcome: Area Under the Plasma Concentration vs Time Curve (AUC) of RGLS8429
Description: Measure area under the plasma concentration vs time curve after RGLS8429 administration
Time Frame: Baseline to Day 15
Reporting Status: Not Posted

6. Secondary Outcome: Amount of RGLS8429 Excreted in Urine
Description: Measure the amount of RGLS8429 excreted in urine after RGLS8429 administration
Time Frame: Baseline to 24-hour
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All Adverse Events were collecting beginning with the start of study drug administration until the Day 29 End of Study Visit.
Arm/Group | RGLS8429, First Dose Level | RGLS8429, Second Dose Level | RGLS8429, Third Dose Level | RGLS8429, Fourth Dose Level | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 3/6 | 1/6 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RGLS8429, First Dose Level (N=6) | RGLS8429, Second Dose Level (N=6) | RGLS8429, Third Dose Level (N=6) | RGLS8429, Fourth Dose Level (N=6) | Matching Placebo (N=8)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT05429073/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT05429073/SAP_001.pdf